CLINICAL TRIAL: NCT02388230
Title: Quantification of Breast RadioTherapy Associated Late Toxicity Using Novel
Brief Title: Quantification of Breast RadioTherapy Associated Late Toxicity Using Novel UltraSound Techniques
Acronym: QuaRTUS
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Royal Marsden NHS Foundation Trust (Other); Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 4220
Record Dates: First submitted 2015-02-20; First posted 2015-03-13 (Estimated); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Breast Radiotherapy Toxicity
Keywords: Breast cancer; Elastography; Ultrasound imaging; Quantification of toxicity; Side-effects
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients 4 or more years post radiotherapy: IMPORT or FAST trial patients who received breast RT previously and are receiving four years (or more) follow-up assessment and have hardening of their breast as a result of breast radiotherapy.
  Interventions: Device: Ultrasound imaging
- Patients 0 to 2 years post breast radiotherapy: Patients who are (1) undergoing, or undergone recently breast RT (general population) and have undergone a clinical assessment either during RT or at 3 month follow-up that found moderate or severe oedema, or (2) IMPORT patients who have received RT and are receiving one or two year follow-up, at which moderate or severe oedema is reported.
  Interventions: Device: Ultrasound imaging

INTERVENTIONS:
Device: Ultrasound imaging

SUMMARY:
Around 20% of women who receive breast radiotherapy (RT) experience moderate to severe breast hardening and shrinkage. These side-effects have been shown to be important factors influencing quality of life after breast radiotherapy. It is thought that the likelihood of developing these side-effects is related to the presence of underlying genetic differences in patients. In order to identify these genetic differences, the severity of side-effects needs to be accurately measured. Currently, clinical assessments are conducted by a clinician but this is not specific enough to be able to relate development of breast shrinkage and hardening to genetic differences. For example, clinical assessment often fails to distinguish between hardness due to swelling (known as oedema) and hardness due to generalised radiation-induced scarring (known as fibrosis). Ultrasound techniques, however, may be able to help quantify and characterise radiotherapy-associated changes in breast tissue allowing for better correlation with genetic abnormalities. Once genetic changes can be identified, adjustment of breast RT treatments (or add drugs) to help reduce side-effects in women at higher genetic risk of side-effects may be possible.

This study tests the ability of two forms of ultrasound, shear-wave elastography (USE) and ultrasound backscatter spectroscopy (UBS), to quantify and characterise breast shrinkage and firmness with a view to using these techniques to measure the late side-effects of breast RT to study the underlying causes of radiotherapy toxicity.

Principle research question: Can a new ultrasound technique (shear wave elastography) measure radiation-induced side-effects in women who have received breast radiotherapy?

ELIGIBILITY:
Inclusion Criteria:

Two patient groups will be included:

1. IMPORT or FAST trial patients who received breast RT previously and have received four (or more) year follow-up assessment which found moderate or severe induration.
2. Patients who are (1) undergoing, or undergone recently, breast RT (general population) and have undergone a clinical assessment that found moderate or severe oedema, or (2) IMPORT HIGH patients who have received RT and have received one or two year follow-up which found moderate or severe oedema.

Exclusion Criteria:

* Patients with bi-lateral breast cancer.
* Patients who have undergone surgery to the contralateral breast for either benign or malignant conditions.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radiotherapy for breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2015-10; Primary Completion 2020-04-08 (Actual); Study Completion 2020-04-08 (Actual)

PRIMARY OUTCOMES:
Young's modulus (kPa) in the irradiated and non-irradiated breast. | Outcome measures will be assessed for each patient during their imaging appointment only. For group 1 patients imaging takes place more than 4 years post radiotherapy, for group 2 patients imaging takes place 3 months to 2 years post radiotherapy.
  Difference in Young's Modulus measured in the irradiated breast and Young's Modulus measured in the non-irradiated breast in patients with reported breast hardness.

CONTACTS AND LOCATIONS:
Overall Officials: Emma J Harris, PhD, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- The Royal Marsden, Sutton, United Kingdom